CLINICAL TRIAL: NCT06999304
Title: Personalized Accelerated Theta Burst Transcardial Magnetic Stimulation in Mild Traumatic Brain Injury
Brief Title: Pilot TMS in Mild TBI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A24-141
Record Dates: First submitted 2025-05-12; First posted 2025-05-31 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Persistent Post Concussive Headache; Mild Traumatic Brain Injury
Keywords: transmagnetic stimulation; functional MRI guided theta burst stimulation; intermittent theta burst stimulation
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Theta burst stimulation (Experimental): There will be a total of 25 theta burst sessions across 5 treatment visits (5 sessions per treatment visit), over a two-week period. Treatment will be applied to 2 brain regions of interest or parcellations: (1) Left 8AV; 2) A personalized region based on imaging and symptom profile.
  Interventions: Device: Intermittent theta burst stimulation

INTERVENTIONS:
Device: Intermittent theta burst stimulation — MagVenture TMS Therapy active coil with theta burst stimulation. Resting motor threshold: 80%; Intermittent theta burst - Number of pulses per session: 1200 pulses; Inter-train interval: 8 seconds; Pulse frequency in burst: 50 Hertz; Continuous theta burst - Number of pulses per session: 1800 pulses; Pulse frequency in burst: 50 Hertz
  Other Names: Transmagnetic stimulation; MagVenture

SUMMARY:
Persistent post-concussive symptoms (PPCS) involve an array of physical, cognitive, and behavioral symptoms lasting more than a month after mild traumatic brain injury (mTBI). 34-44% of people with mTBI or concussion present with a considerable burden of PPCS 3-6 months after injury. There is currently no standardized treatment for PPCS, nor FDA approved medication for any neuropsychiatric or neurocognitive symptoms associated with mTBI. Transcranial magnetic stimulation (TMS) shows promise as a treatment for PPCS; however, the current one-size-fits-all approach does not address the heterogeneity of symptoms. We propose utilization of resting state functional MRI (rs-fMRI) guided rTMS to target personalized brain networks burdened with PPCS.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of mTBI at least 4 weeks prior but not exceeding 12 months prior to the time of screening
2. Age 18-65 years at the time of mTBI
3. High burden of post concussive symptoms at time of screening, as measured by symptoms questionnaire (PCSS) ≥35*

Exclusion Criteria:

1. Inability to tolerate imaging; contraindication of imaging due to implants or metal
2. Seizure disorder, active alcohol or substance use disorder
3. Inability to speak and read English
4. Anything else that, in the opinion of the PI/study physician, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.
5. Subject is pregnant or breast feeding
6. Subject has participated in a clinical interventional trial in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with anomalous parcellations - developing the method of personalization of TMS for PPCS | baseline
  Percentage of participants matched with anomalous parcellations based on one of the 2 top ranked burdensome symptoms/symptom profile. If an anomalous parcellation matching one of the top 2 ranked symptom profiles can be identified in at least 16 out of 20 (80%) of participants, the trial will be considered a success.
Anomalous parcellations - developing the method of personalization of TMS targets for PPCS | baseline
  Names and number of anomalous parcellations identified using connectivity analysis and targets available to treat with TMS based on symptom profiles
Distribution of complaints for PPCS | baseline
  Distribution of chief symptom/complaints among participants measured by concussion clinical profile (CP) screen
Mapping of complaints to anomalous parcellations | baseline
  Mapping of chief symptom/complaints to parcellations based on literature and connective abnormalities

SECONDARY OUTCOMES:
Feasibility - rate of completed treatment | 4 weeks
  Percent of participants who complete 4 out of the 5 treatment visits.
Fidelity | 4 weeks
  Percent of participants who complete all sessions of treatment.
Safety - adverse events | 16 weeks
  Frequency of each adverse events.
Acceptability | 4 weeks
  This survey will be used to understand the subject's experience with TMS and whether they feel it is an acceptable form of treatment. Questions will be both open-ended and quantitative (Likert scale). In this study, participants will be asked about their level of satisfaction with various aspects of the treatment. This survey is not standardized. Scores presented as percent of subject responses. Range: [0-100]. Higher percentage indicates more acceptability to this form of treatment.

OTHER OUTCOMES:
Explore pre-post changes concurrent with personalized TMS on PPCS - global post-concussion scale | baseline, 1 week post-treatment, 4 week post-treatment, 12 week post-treatment
  Pre-post change in global post-concussion scale - Rivermead Post-Concussion Symptoms Questionnaire (RPQ) from baseline to 4- and 12-weeks post-enrollment. The RPQ consists of 16 questions about symptoms experienced after a head injury, rated on a scale of 0-4. Range [0-64]. A higher score indicates more severe symptoms. A positive change from pre to post (post score-pre score=change) indicates that symptoms get worse.
Explore pre-post changes concurrent with personalized TMS on PPCS - generalized anxiety | baseline, 1 week post-treatment, 4 week post-treatment, 12 week post-treatment
  Pre-post change in symptom specific profile scale (general anxiety disorder-7 (GAD7)) from baseline to 4- and 12-weeks post-enrollment. The GAD7 is a 7-item anxiety scale that is self-administered, valid, and an efficient tool for screening for GAD and assessing its severity in clinical practice and research. Range: [0-21] A higher score indicates more anxiety. A positive change from pre to post (post score-pre score=change) indicates that anxiety symptoms get worse.
Explore pre-post changes concurrent with personalized TMS on PPCS - speed of forgetting | baseline, 1 week post-treatment, 4 week post-treatment, 12 week post-treatment
  Pre-post change in symptom specific profile scale (speed of forgetting (SoF)) from baseline to 4- and 12-weeks post-enrollment. The SOF quantifies the rate of episodic trace decay without the effects of learning. Content is presented as cue-pair associates and assessed through multiple-choice or verbal recall questions. This test is 8 minutes long.
  Range: [0-1]. A higher score indicates more memory impairment. A positive change from pre to post (post score-pre score=change) indicates that memory gets worse.
Explore pre-post changes concurrent with personalized TMS on PPCS - CP screen | baseline, 1 week post-treatment, 4 week post-treatment, 12 week post-treatment
  Pre-post change in Concussion Clinical Profiles Screening (CP) from baseline to 4- and 12-weeks post-enrollment. The CP is a 29 item self report tool to assess clinical profiles associated with concussion. Range: [0-87]. A higher score indicates more severe symptoms. A positive change from pre to post (post score-pre score=change) indicates that symptoms get worse.
Explore pre-post changes concurrent with personalized TMS on PPCS - respond to treatment | baseline, 1 week post-treatment, 4 week post-treatment, 12 week post-treatment
  Percent of participants that respond to treatment based on improvement in symptom specific scales at 1- 4- and 12-weeks post-enrollment, defined as either show minimally clinically important difference (MCID) ≥2 SD improvement from baseline at a given timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Kashyap, MBBS, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be shared with other researchers.